CLINICAL TRIAL: NCT06355167
Title: Interventional, Open-label Study of the Effect of an Aquaporin-1 Inhibitor, the Bacopaside II Contained in Bacopa-400® , on Oxidative Stress in Healthy Volunteers: BacOxy_I Study
Brief Title: Effect of Oral Intake of Bacopa Monneiri on Vascular Oxidative Stress
Acronym: Bacoxy_I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Montiel Virginie, Head of the intensive care unit, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Bacoxy_I
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Oxidative Stress; Cardiovascular Diseases; Bacopaside II; Bacopa Monnieri; Endothelial Dysfunction; Aquaporin 1; AQP1
Keywords: vascular oxidative stress; aquaporin 1; AQP1; hydrogen peroxide; cardiovascular diseases; Bacopa monnieri; Bacopaside II; endothelial dysfunction
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Group A (n=10): 400mg/d of Bacopa monnieri Broup B (n=10): 800 mg/d of Bacopa monnieri
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 dose: 1 capsule of Bacopa monnieri (400mg) (Other): Group A: 400mg/d of Bacopa monnieri
  Interventions: Dietary Supplement: Bacopa monnieri
- 2 doses: 2 capsules of Bacopa monnieri (800mg) (Other): Group B: 800 mg/d of Bacopa monnieri
  Interventions: Dietary Supplement: Bacopa monnieri

INTERVENTIONS:
Dietary Supplement: Bacopa monnieri — Daily oral intake of Bacopa monnieri during 6 weeks
  Other Names: Bacopa-400

SUMMARY:
Bacoxy_I study aims to evaluate the efficacy of a standardized Bacopa monnieri extract, Bacopa-400®, on vascular oxidative stress.

DETAILED DESCRIPTION:
The Bacopa-400® is a standardized extract of a plant called Bacopa Monnieri, which mainly grows in India and neighboring countries. The virtues of this plant, also called Brahmi, have been used in Ayurvedic medicine for millennia in the treatment of chronic neurological diseases accompanied by cognitive impairment and memory disorders, as well as for stress management. Several companies have subsequently improved the preparation of standardized extracts of Bacopa Monnieri. Bacopa-400® from the Belgian firm Deba Pharma™ was selected because it adheres to good manufacturing practices (GMP). Currently, there are over 289 studies listed regarding the positive role of Bacopa monnieri in cognitive functions in both young and elderly subjects. Furthermore, no major side effects have been reported following the use of this plant extract in acute or chronic administration in hundreds of people of all ages.

Bacopa monnieri plant contains several bacosides, including the Bacopaside II a specific inhibitor of the water channel Aquaporin 1 (AQP1). AQP1 is part of the aquaporin family responsible for bidirectional transmembrane water transport. It is the most abundant aquaporin in mammalian cardiovascular tissue, present in myocardial cells, endothelial cells, and red blood cells. AQP1, more than a water channel, is also a peroxiporin able to facilitate the passage of hydrogen peroxide (H2O2), involved in oxidative stress.

In previous work, the Pharmacology and Therapeutics (FATH) department from UCLouvain (Brussels) discovered the protective effect of Bacopaside II on cardiovascular oxidative stress. Through a series of experiments, it was demonstrated that Bacopaside II dose dependently attenuates the passage of H2O2 into cardiac myocytes, thus preventing hypertrophy induced by neurohormones. Additionally, in murine models, oral administration of Bacopa monnieri extract attenuated cardiac hypertrophy triggered by hypertrophic stimuli. This cardiac protection occurs through inhibition of AQP1.

Based on this premises, a clinical investigation was undertaken to explore the potential of Bacopa-400® in attenuating vascular oxidative stress among healthy volunteers. This interventional, open-label and monocentric comprised two groups. Group A received a daily dose of 400 mg and Group B a daily dose of 800 mg over a 6-week period, followed by a 4-week observation period after the cessation of treatment.

The primary objective of this study was to assess the impact of Bacopa-400® on oxidative stress in healthy individuals and determine the optimal dosage for maximal efficacy. Furthermore, the study analyzed the incidence, severity, and frequency of adverse events, including suspected unexpected serious adverse events (SUSAR).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Effective contraception

Exclusion Criteria:

* Any chronic disease
* Any chronic use of drug
* Pregnancy and breast feeding
* Gastro-intestinal diseases (e.g. ulcer, gastro-oesophageal reflux, lactose intolerance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Ex vivo DCFDA test on red blood cells (RBCs) | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  DCFA (dichlorofluorescein diacetate) is a probe used to assess the presence of intracellular reactive oxygen species (ROS). Red blood cells are incubated with DCFA and extracellular hydrogen peroxide (H2O2). After passive diffusion into the cells and upon encountering ROS, DCFDA undergoes conversion to produce a highly fluorescent compound, the DCF (2',7'-Dichlorofluorescein). This resulting fluorescence intensity (arbitrary unit) was quantified using FACS. This technique allowed us to measure kinetically the entry of ROS as H2O2 in RBCs.
Plasma lipid peroxydes | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Lipid peroxidation (µM) is a form of oxidative damage that impacts cellular membranes, lipoproteins, and other lipid-containing molecules under conditions of oxidative stress. Assessing changes in lipid peroxide levels during the study served as a reflection of oxidative status. Plasma lipid peroxides were quantified using a colorimetric test using the 3,3',5,5'-tetramethylbenzidine (TMB).
Methemoglobin in red blood cells | Baseline (V0), 6 weeks (V4), 10 weeks (V6)
  Methemoglobin is the oxidized form of hemoglobin, where the iron atom in the heme group is oxidized from the ferrous to the ferric state. Exposure to oxidative stress can lead to the formation of methemoglobin making the latter a biomarker of vascular oxidative stress. Methemoglobin levels (arbitrary unit) were measured by electron paramagnetic resonance spectroscopy.
Nitrosylated hemoglobin (HbNO) in red blood cells | Baseline (V0), 6 weeks (V4), 10 weeks (V6)
  Vascular oxidative stress is involved in the decreased of nitric oxide (NO) bioavailability. Erythrocyte 5-α-coordinate nitrosyl-hemoglobin or nitrosylated hemoglobin (HbNO) is a complexe between NO and deoxyhemoglobin serving as a marker for NO bioavailability. HbNO levels (nM) were quantified using electron paramagnetic resonance spectroscopy

SECONDARY OUTCOMES:
haemoglobin | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  The haemoglobin (g/L) is part of hemogram, a quantitative and qualitative analysis of blood constituents. This test was performed to reiterate the known safety of Bacopa monnieri on the systemic circulation after oral ingestion.
haematocrit | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  The haematocrit (g/L) is part of hemogram, a quantitative and qualitative analysis of blood constituents. This test was performed to reiterate the known safety of Bacopa monnieri on the systemic circulation after oral ingestion.
Red blood cells count | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  The red blood cells count (10^6/µL) is part of hemogram, a quantitative and qualitative analysis of blood constituents. This test was performed to reiterate the known safety of Bacopa monnieri on the systemic circulation after oral ingestion.
Sodium | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Sodium (mM) is part of ion count. Electrolyte concentrations were evaluated to monitor the impact of Bacopa monnieri's diuretic effect on blood ion levels.
Potassium | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Potassium (mM) is part of ion count. Electrolyte concentrations were evaluated to monitor the impact of Bacopa monnieri's diuretic effect on blood ion levels.
Bicarbonate | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Bicarbonate (mM) is part of ion count. Electrolyte concentrations were evaluated to monitor the impact of Bacopa monnieri's diuretic effect on blood ion levels.
Total cholesterol | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Total cholesterol (mg/dL) is part of the lipogram, to assess the effect of oral intake of Bacopa monnieri on the lipid metabolism.
High-Density Lipoprotein (HDL) cholesterol | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  HDL cholesterol (mg/dL), is part of the lipogram, to assess the effect of oral intake of Bacopa monnieri on the lipid metabolism.
Low-Density Lipoprotein (LDL) cholesterol | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  LDL cholesterol (mg/dL) is part of the lipogram, to assess the effect of oral intake of Bacopa monnieri on the lipid metabolism.
Triglycerides | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Triglycerides (mg/dL) is part of the lipogram, to assess the effect of oral intake of Bacopa monnieri on the lipid metabolism.
aspartate aminotransferase (ASAT), (U/L) | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  ASAT (U/L) was assessed to evaluate the safety of Bacopa monnieri on liver function following oral intake.
alanine aminotransferase (ALAT) (U/L) | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  ALAT (U/L) was assessed to evaluate the safety of Bacopa monnieri on liver function following oral intake.
gamma-glutamyl-transferase (GGT) level | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  GGT (U/L) was assessed to evaluate the safety of Bacopa monnieri on liver function following oral intake
Creatinine | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Creatinine (mg/dl) was measured to assess the impact of oral intake of Bacopa monnieri on renal function.
Glomerular filtration rate | Baseline (V0), 2 weeks (V2), 6 weeks (V4), 10 weeks (V6)
  Glomerular filtration rate (ml/min/m²) was measured to assess the impact of oral intake of Bacopa monnieri on renal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique universitaires saint luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montiel V, Bella R, Michel LYM, Esfahani H, De Mulder D, Robinson EL, Deglasse JP, Tiburcy M, Chow PH, Jonas JC, Gilon P, Steinhorn B, Michel T, Beauloye C, Bertrand L, Farah C, Dei Zotti F, Debaix H, Bouzin C, Brusa D, Horman S, Vanoverschelde JL, Bergmann O, Gilis D, Rooman M, Ghigo A, Geninatti-Crich S, Yool A, Zimmermann WH, Roderick HL, Devuyst O, Balligand JL. Inhibition of aquaporin-1 prevents myocardial remodeling by blocking the transmembrane transport of hydrogen peroxide. Sci Transl Med. 2020 Oct 7;12(564):eaay2176. doi: 10.1126/scitranslmed.aay2176. PMID 33028705
- [Background] Montiel V, Leon Gomez E, Bouzin C, Esfahani H, Romero Perez M, Lobysheva I, Devuyst O, Dessy C, Balligand JL. Genetic deletion of aquaporin-1 results in microcardia and low blood pressure in mouse with intact nitric oxide-dependent relaxation, but enhanced prostanoids-dependent relaxation. Pflugers Arch. 2014 Feb;466(2):237-51. doi: 10.1007/s00424-013-1325-x. Epub 2013 Jul 20. PMID 23873354
- [Background] Pravina K, Ravindra KR, Goudar KS, Vinod DR, Joshua AJ, Wasim P, Venkateshwarlu K, Saxena VS, Amit A. Safety evaluation of BacoMind in healthy volunteers: a phase I study. Phytomedicine. 2007 May;14(5):301-8. doi: 10.1016/j.phymed.2007.03.010. Epub 2007 Apr 17. PMID 17442556
- [Background] Stough C, Downey LA, Lloyd J, Silber B, Redman S, Hutchison C, Wesnes K, Nathan PJ. Examining the nootropic effects of a special extract of Bacopa monniera on human cognitive functioning: 90 day double-blind placebo-controlled randomized trial. Phytother Res. 2008 Dec;22(12):1629-34. doi: 10.1002/ptr.2537. PMID 18683852
- [Background] Dave UP, Dingankar SR, Saxena VS, Joseph JA, Bethapudi B, Agarwal A, Kudiganti V. An open-label study to elucidate the effects of standardized Bacopa monnieri extract in the management of symptoms of attention-deficit hyperactivity disorder in children. Adv Mind Body Med. 2014 Spring;28(2):10-5. PMID 24682000